CLINICAL TRIAL: NCT01766219
Title: A Pilot Open-Label Clinical Trial of CPI-613 in Patients With Advanced Bile Duct Cancers
Brief Title: CPI-613 in Treating Patients With Advanced or Metastatic Bile Duct Cancer That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB00022533; NCI-2013-00063 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH); CCCWFU 59212 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2013-01-10; First posted 2013-01-11 (Estimated); Results first posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-04

CONDITIONS: Adult Primary Cholangiocellular Carcinoma; Advanced Adult Primary Liver Cancer; Cholangiocarcinoma of the Extrahepatic Bile Duct; Cholangiocarcinoma of the Gallbladder; Localized Unresectable Adult Primary Liver Cancer; Metastatic Extrahepatic Bile Duct Cancer; Recurrent Adult Primary Liver Cancer; Recurrent Extrahepatic Bile Duct Cancer; Unresectable Extrahepatic Bile Duct Cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Carcinoma, Hepatocellular | interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: (6,8-bis[benzylthio]octanoic acid) 2,300 mg/m² (Experimental): Participants will not be treated with CPI-613 during pre-Cycle 1 and will only be treated with 3 weeks on/1 week off at 2,300 mg/m² as a starting dose. If none of these 3 participants develop a dose-limiting toxicity through Cycle 1, the dose for the 3-weeks-on-1-week-off treatment cycles will be 3,000 mg/m² in all subsequent participants in this trial.
  Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1 and 4 of weeks 1-3. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive up to 4 more courses of treatment.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid
- Arm 2: (6,8-bis[benzylthio]octanoic acid) 1,200/3,00 mg/m² (Experimental): Participants will received pre-cycle 1 week dose at 1200 mg/m² and dosing will escalate to 3,000 mg/m² for the three weeks on, one week off cycle.
  Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1 and 4 of weeks 1-3. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive up to 4 more courses of treatment.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid
- Arm 3 (6,8-bis[benzylthio]octanoic acid) 600/3,000 mg/m² (Experimental): Participants will received pre-cycle 1 week dose at 600 mg/m² and dosing will escalate to 3,000 mg/m² for the three weeks on, one week off cycle.
  Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1 and 4 of weeks 1-3. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive up to 4 more courses of treatment.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid

INTERVENTIONS:
Drug: 6,8-bis(benzylthio)octanoic acid — Given IV
  Other Names: alpha-lipoic acid analogue CPI-613; CPI-613

SUMMARY:
This pilot clinical trial studies 6,8-bis(benzylthio)octanoic acid in treating patients with advanced or metastatic cholangiocarcinoma that cannot be removed by surgery. 6,8-Bis(benzylthio)octanoic acid may stop the growth of cholangiocarcinoma by blocking blood flow to the tumor

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and efficacy of CPI-613 (6,8-bis[benzylthio]octanoic acid) in patients with advanced unresectable cholangiocarcinoma who have failed available therapies.

OUTLINE:

Pre-cycle: Patients receive 6,8-bis(benzylthio)octanoic acid intravenously (IV) over 2 hours on days 1-5, 1 week prior to course 1.

Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1 and 4 of weeks 1-3. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive up to 4 more courses of treatment.

After completion of study treatment, patients are followed up bimonthly.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and cytologically proven cholangiocarcinoma of any type (including intrahepatic cholangiocarcinoma, extrahepatic primary cholangiocarcinoma, hilar cholangiocarcinomas, cholangiocarcinomas located in the gall bladder or hepatic capsule effraction, and carcinoma of the Ampulla of Vater, etc.) that is not amenable to surgery, radiation, or combined modality therapy with curative intent, and has failed or is not eligible for available chemotherapies such as gemcitabine with or without platinum
* Local, locally-advanced, or metastatic disease documented as having shown progression on a scan (e.g., computed tomography [CT], magnetic resonance imaging [MRI])
* Measurable tumor according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria with at least one unidimensionally measurable target lesion
* No evidence of biliary duct obstruction, unless obstruction is controlled by local treatment or, in whom the biliary tree can be decompressed by endoscopic or percutaneous stenting with subsequent reduction in bilirubin to below 1.5 x upper level of normal (ULN)
* No acute toxic effects from previous treatment superior to grade 1 at the start of the study
* Eastern Cooperative Oncology Group (ECOG) performance status being 0-3
* Expected survival > 3 months
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists
* Granulocyte count >= 1500/mm^3
* White blood cell (WBC) >= 3500 cells/mm^3 or >= 3.5 bil/L
* Platelet count >=100,000 cells/mm^3 or >=100 bil/L
* Absolute neutrophil count (ANC) >=1500 cells/mm^3 or >=1.5 bil/L
* Hemoglobin >= 9 g/dL or >= 90 g/L
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x upper normal limit (UNL), alanine aminotransferase (ALT/serum glutamate pyruvate transaminase [SGPT]) =< 3 x UNL (=< 5 x UNL if liver metastases present)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 2.0 mg/dL or 177 µmol/L
* International normalized ratio or INR must be =< 1.5
* No evidence of active infection and no serious infection within the past month
* Mentally competent, ability to understand and willingness to sign the informed consent form

Exclusion Criteria:

* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 2 weeks prior to initiation of CPI-613 treatment
* Serious medical illness that would potentially increase patients' risk for toxicity
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease)
* Pregnant women, or women of child-bearing potential not using reliable means of contraception (because the teratogenic potential of CPI-613 is unknown)
* Lactating females
* Fertile men unwilling to practice contraceptive methods during the study period
* Life expectancy less than 3 months
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Unwilling or unable to follow protocol requirements
* Dyspnea with moderate exertion; patients with clinically significant pleural or pericardial effusions
* Active heart disease including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, symptomatic myocardial infarction, or symptomatic congestive heart failure; also patients with a history of myocardial infarction that is < 1 year prior to registration, or patients with previous congestive heart failure (< 1 year prior to registration) requiring pharmacologic support or with left ventricular ejection fraction < 50%)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome)
* Evidence of active infection, or serious infection within the past month
* Patients with known human immunodeficiency virus (HIV) infection
* Patients who have received cancer immunotherapy of any type within the past 2 weeks prior to initiation of CPI-613 treatment
* Requirement for immediate palliative treatment of any kind including surgery
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months
* Prior illicit drug addiction
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-05; Primary Completion 2018-04 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caio Rocha Lima, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m²: Patients receive 6,8-bis(benzylthio)octanoic acid IVover 2 hours on days 1 and 4 of weeks 1-3. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive up to 4 more courses of treatment.
  6,8-bis(benzylthio)octanoic acid: Given IV
- Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m²: Pre-cycle: Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5, 1 week prior to course 1.
  Patients receive 6,8-bis(benzylthio)octanoic acid IVover 2 hours on days 1 and 4 of weeks 1-3. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive up to 4 more courses of treatment.
  6,8-bis(benzylthio)octanoic acid: Given IV
- Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m²: Pre-cycle: Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5, 1 week prior to course 1.
  Patients receive 6,8-bis(benzylthio)octanoic acid IVover 2 hours on days 1 and 4 of weeks 1-3. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive up to 4 more courses of treatment.
Period: Overall Study
Arm/Group | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m²
Started | 4 | 2 | 11
Completed | 4 | 2 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m²: Pre-cycle: Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5, 1 week prior to course 1.
  Patients receive 6,8-bis(benzylthio)octanoic acid IVover 2 hours on days 1 and 4 of weeks 1-3. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive up to 4 more courses of treatment.
  6,8-bis(benzylthio)octanoic acid: Given IV
- Total: Total of all reporting groups
Arm/Group | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m² | Total
Number analyzed (Participants) | 4 | 2 | 11 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 6 | 11
  >=65 years | 0 | 1 | 5 | 6
Age, Continuous [Mean (Full Range); unit: years] | 52 [47 to 61] | 66 [56 to 75] | 62 [48 to 78] | 57 [47 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 9
  Male | 1 | 0 | 7 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 2 | 11 | 17
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 4 | 2 | 9 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Estimated using Kaplan-Meier techniques.
Time Frame: From the first dose of 6,8-bis(benzylthio)octanoic acid to death, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m²
Number analyzed (Participants) | 4 | 2 | 11
months | 4.7 [3.2 to 11.0] | 1.6 [0.95 to 2.3] | 3.94 [2.4 to 8.4]

2. Secondary Outcome: Response Rate Defined as Proportion of Patients With Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD)
Description: Using the RECIST version 1.1 as defined by patient with 95% confidence interval will be included. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:the appearance of one or more new lesions is also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: From the start of the treatment until disease progression, assessed up to 4 year
Measure: Number; unit: participants
Groups:
- Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m²; Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m²; Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m²: Pre-cycle: Patients receive 6,8-bis(benzylthio)octanoic acid IV over 2 hours on days 1-5, 1 week prior to course 1.
  Patients receive 6,8-bis(benzylthio)octanoic acid IVover 2 hours on days 1 and 4 of weeks 1-3. Treatment repeats every 4 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity. Patients responding to treatment may receive up to 4 more courses of treatment.
  6,8-bis(benzylthio)octanoic acid: Given IV
Arm/Group | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m²
Number analyzed (Participants) | 4 | 2 | 11
participants
  Stable Disease | 0 | 2 | 2
  Progression | 4 | 0 | 7
  Not Evaluable | 0 | 0 | 2

3. Secondary Outcome: Progression-free Survival
Description: Estimated using Kaplan-Meier techniques as well as RECIST 1.1. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note:the appearance of one or more new lesions is also considered progression).
Time Frame: From the first dose of 6,8-bis(benzylthio)octanoic acid to disease progression (DP) or death due to any cause, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m²
Number analyzed (Participants) | 4 | 2 | 11
months | 1.6 [1.1 to 3.8] | 0 [NA to NA] — Both participants in Arm 2 progressed at the exact same time, the statistician couldn't get a median and a confidence interval. A mean or 0.5589 and standard deviation of 0 was reported | 2.5 [1.4 to 3.6]

4. Secondary Outcome: Number of Participants With Adverse Events Using the National Cancer Institute Common Terminology Criteria
Description: Adverse events will be captured using the National Cancer Institute Common Terminology Criteria (NCI CTCAE) version 3.0
Time Frame: Up to 1 month completion of study treatment, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m²
Number analyzed (Participants) | 4 | 2 | 11
Participants | 4 | 2 | 11

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: All-Cause Mortality data, serious Adverse Events and Other (Not Including Serious) Adverse Events data were collected for 17 participants.
Arm/Group | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m² | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m²
All-Cause Mortality (participants affected / at risk) | 4/4 | 2/2 | 11/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/2 | 1/11
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m² (N=4) | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m² (N=2) | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m² (N=11)
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 (1) | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1)
Hypotension (Vascular disorders) | 0 | 0 | 1 (1)
Sepsis (Infections and infestations) | 0 | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 2,300 mg/m² (N=4) | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 1,200/3,000 mg/m² (N=2) | Treatment (6,8-bis[Benzylthio]Octanoic Acid) 600/3,000 mg/m² (N=11)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 1 (1) | 4 (4)
Alanine amniotransferase increased (Investigations) | 1 (1) | 0 (0) | 7 (7)
Alkaline phosphastase increased (Investigations) | 4 (4) | 1 (1) | 11 (11)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 8 (8)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1) | 7 (7)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 1 (1) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (3) | 0 (0) | 6 (6)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 2 (2) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 5 (5)
Fatigue (General disorders) | 3 (3) | 1 (1) | 9 (9)
GGT increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cystic duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 6 (6)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2) | 9 (9)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 7 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4)
Lymphocyte count decreased (Investigations) | 3 (3) | 0 (0) | 11 (11)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 8 (8)
Pancreas infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 5 (5)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 6 (6)
White blood count decreased (Investigations) | 2 (2) | 0 (0) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 5 (5)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 7 (7)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 2 (2)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 9 (9)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Edema face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diffuse abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 5 (5)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3)
Esophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatic duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Iron elevated (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) — Iron level at 41
Muscle weakness, left side (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness, right side (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness, lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness, trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness, upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
General body aches (General disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders Other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — Patient was not confused but "spacey"
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased concentration (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Erythema, left extremity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechia, right buttock (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Close to eye
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
[Not specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT01766219/Prot_SAP_000.pdf